CLINICAL TRIAL: NCT01642758
Title: An Open-Label Phase 2 Study of HQK-1001 in Subjects With Beta Thalassemia Intermedia
Brief Title: Trial of HQK-1001 in Beta Thalassemia Intermedia in Lebanon
Acronym: LB-04-THAL
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Boston University (Other)
Collaborators: HemaQuest Pharmaceuticals Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HQK-P2-THAL
Record Dates: First submitted 2012-07-12; First posted 2012-07-17 (Estimated); Last update posted 2013-03-14 (Estimated); Status verified 2013-03

CONDITIONS: Beta Thalassemia Intermedia
Keywords: Thalassemia intermedia; Fetal hemoglobin; Hemoglobin
MeSH Terms: conditions — beta-Thalassemia | interventions — 2,2-dimethylbutyric acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Sodium 2,2 dimethylbutyrate (Experimental): A single dose (20 mg/kg/day) of study drug will be taken once per day by mouth.
  Interventions: Drug: Sodium 2,2 dimethylbutyrate

INTERVENTIONS:
Drug: Sodium 2,2 dimethylbutyrate — Oral capsules, dose 20 mg/kg/day, once per day for 26 weeks
  Other Names: ST20

SUMMARY:
Beta thalassemia intermedia syndromes are genetic anemias caused by mutations which reduce production of beta globin, a major component of adult hemoglobin A, the protein which delivers oxygen throughout the body. Patients suffer from poor growth, fatigue, heart failure, endocrine deficiencies, and eventually, many require chronic blood transfusions. There is no approved therapeutic for the deficiency of beta globin chains in beta thalassemia.

This trial will study an oral therapeutic which stimulates production of fetal globin, an alternate type which is produced by all humans, but is normally switched off in infancy. This type of globin can compensate for the missing protein in beta thalassemia.

DETAILED DESCRIPTION:
This is a trial of an experimental oral medicine which stimulates production of fetal hemoglobin, an innate type of hemoglobin which is normally made but is suppressed in infancy. Fetal globin (HbF) can perform the function of the missing beta globin and reduce anemia in beta thalassemia, when it is produced in higher amounts than normal.

In this trial, 10 patients with beta thalassemia intermedia in Lebanon will all receive the study drug for 6 months at a dose which has been previously shown to be safe in normal volunteers and in beta thalassemia and sickle cell patients and to stimulate fetal globin production in many, when given for brief periods. The purpose of this trial is the following:

1. To determine if total hemoglobin levels increase above baseline in some subjects when the study drug is taken for 26 weeks.
2. To determine if fetal globin is increased above baseline levels in a proportion of subjects when the study drug is taken for 26 weeks.
3. To determine the number of adverse events which occur with 26 weeks of administration of the study drug in beta thalassemia intermedia subjects.

After a screening period, the subjects will take the study drug at home once a day. They will be seen once every 4 weeks for examinations and laboratory tests during the dosing period and for 4 weeks afterwards.

This trial will provide an important step in evaluating a potential treatment for patients with beta thalassemia intermedia, that can be used around the world, if it is effective and safe.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of beta thalassemia intermedia
* Ages 16-50 years
* Average total Hgb levels between 6.0 and 9.0 gm/dl within 30 days of initial dose of study drug
* Able to comply with all study procedures
* If female and of childbearing potential, must have a documented negative pregnancy test prior to entry and every 4 weeks

Exclusion Criteria:

* Red blood cell transfusions within 3 months prior to administration of study drug
* QT Segment corrected (QTc)> 450 msec
* Use of Erythropoiesis Stimulating Agents(ESAs)within 9 days of first dose
* Hydroxyurea treatment within 6 months of first study drug
* History of significant arrythmias, syncope, or resuscitation
* Alanine Transaminase (ALT)> 4x upper limit of normal
* Serum creatinine > 1.5 mg/dl
* Sse of iron chelating agents within 7 days of first dose
* Pulmonary hypertension requiring oxygen therapy

Ages: 16 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 10 (Actual)
Dates: Start 2012-05; Primary Completion 2012-11 (Actual); Study Completion 2013-01 (Actual)

PRIMARY OUTCOMES:
To measure changes from baseline in total hemoglobin when HQK-1001 is administered orally for 26 weeks in subjects with beta thalassemia intermedia. | 6 months
  Baseline hemoglobin levels will be determined in each subject and averaged from levels obtained on a screening visit and on day one of the study, before any drug is taken. Hemoglobin levels will then be analyzed every 4 weeks during 26 weeks of taking the study drug and for 4 weeks after the dosing is completed. Changes from baseline will be determined.

SECONDARY OUTCOMES:
To measure the number of adverse events which occur with HQK-1001 treatment when given over 26 weeks in beta thalassemia intermedia. | 6 months
  Adverse events which occur during HQK-1001 administration for 26 weeks will be recorded every 4 weeks.
To measure changes from baseline in HbF during treatment with HQK-1001 for 26 weeks in beta thalassemia intermedia. | 6 months
  Levels of HbF will be averaged from a screening visit and day 1 of the study, prior to any drug treatment. HbF levels will then be measured every 4 weeks during treatment and for 4 weeks after the treatment, and compared to each subject's baseline value. The number of subjects in which an increase in HbF develops above individuals' average baseline value will be obtained.

CONTACTS AND LOCATIONS:
Overall Officials: Susan P Perrine, MD, Study Director — Boston University; Adlette Inati, MD, Principal Investigator — Chronic Care Center and Rafik Hariri University Hospital, Beirut, Lebanon
Locations (1):
- Chronic Care Center, Beirut, Lebanon

REFERENCES:
- [Background] Perrine SP, Wargin WA, Boosalis MS, Wallis WJ, Case S, Keefer JR, Faller DV, Welch WC, Berenson RJ. Evaluation of safety and pharmacokinetics of sodium 2,2 dimethylbutyrate, a novel short chain fatty acid derivative, in a phase 1, double-blind, placebo-controlled, single-dose, and repeat-dose studies in healthy volunteers. J Clin Pharmacol. 2011 Aug;51(8):1186-94. doi: 10.1177/0091270010379810. Epub 2011 Mar 21. PMID 21422239
- [Background] Perrine SP, Castaneda SA, Chui DH, Faller DV, Berenson RJ, Siritanaratku N, Fucharoen S. Fetal globin gene inducers: novel agents and new potential. Ann N Y Acad Sci. 2010 Aug;1202:158-64. doi: 10.1111/j.1749-6632.2010.05593.x. PMID 20712788